CLINICAL TRIAL: NCT00804817
Title: Somatic-psychosocial Multidisciplinary Care Concept for Oncologic Patients Undergoing Hematopoietic Stem Cell Transplantation (HSCT): a Prospective Non-randomized Clinical Trial
Brief Title: Somatic-psychosocial Care Concept for Oncologic Patients Undergoing Hematopoietic Stem Cell Transplantation (HSCT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Collaborators: Deutsche Krebshilfe e.V., Bonn (Germany) (Other)
Responsible Party: Margarete Landenberger, Prof. PhD, Martin-Luther-University Halle-Wittenberg, Medical Faculty, Department for Health and Nursing Science
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: DKH-Project; DKH Grand Nr. 107498
Record Dates: First submitted 2008-12-08; First posted 2008-12-09 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2008-12

CONDITIONS: Oral Mucositis; Malnutrition
Keywords: self management; adherence; activity enhancement; oral mucositis prevention; and mal nutrition prevention; cancer; hematopoietic stem cell transplantation (HSCT); loss of activity
MeSH Terms: conditions — Stomatitis; Malnutrition; Neoplasms | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Care as usual (Active Comparator): Care as usual, i.e. standard physical activity enhancement, oral mucositis prevention and treatment and mal nutrition prevention
  Interventions: Behavioral: Control Group
- SCION-HSCT program (Experimental): Patients receive SCION-HSCT program a multi-modular somatic-psycho-social care intervention. consisting of 3 modules: Activity Enhancement, Oral Mucositis Prevention and Mal-Nutrition Avoidance.
  The intervention will be conducted by specially trained oncology nurses and will include components of knowledge, skills training, and coaching to improve self management. The intervention starts at admission followed by booster sessions during the period of hospitalization. Patients will be scheduled to an individualized physical activity program incl. endurance training on light level 60-80% of max heart rate. Additionally the patient will be counselled to follow a mouth care protocol based on self assessment of the mouth to prevent oral mucositis. Both interventions are accompanied by a systematic screening of the nutritional situation. All three interventions are aimed to improve patients' adherence to self management strategies of side effects.
  Interventions: Behavioral: SCION-HSCT program

INTERVENTIONS:
Behavioral: Control Group — Control: Care as usual, i.e. standard physical activity enhancement, oral mucositis prevention and treatment and mal nutrition prevention
  Arms: Care as usual
Behavioral: SCION-HSCT program — Intervention: Patients receive SCION-HSCT program a multi-modular somatic-psycho-social care intervention. consisting of 3 modules: Activity Enhancement, Oral Mucositis Prevention and Mal-Nutrition Avoidance.
  The intervention will be conducted by specially trained oncology nurses and will include components of knowledge, skills training, and coaching to improve self management. The intervention starts at admission followed by booster sessions during the period of hospitalization. Patients will be scheduled to an individualized physical activity program incl. endurance training on light level 60-80% of max heart rate. Additionally the patient will be counselled to follow a mouth care protocol based on self assessment of the mouth to prevent oral mucositis. Both interventions are accompanied by a systematic screening of the nutritional situation. All three interventions are aimed to improve patients' adherence to self management strategies of side effects.
  Arms: SCION-HSCT program

SUMMARY:
This study will test the SCION (Self care improvement through oncology nursing)-HSCT program a multi-modular, somatic-psycho-social care intervention to improve self management in oncologic patients undergoing HSCT. The study will determine if the self management skills of the patients to enhance:

* physical activity,
* prevention of oral mucositis and
* mal nutrition during the period of hospitalization.

It is hypothesized that patients who receive the multi-modular somatic-psycho-social care intervention will have better health related quality of life (HRQoL).

DETAILED DESCRIPTION:
According to Precede Model of health behavior from Green - modified by our research group - patients self management skills are affected by the patients' knowledge, activities and attitude to self management.

Therefore, we propose a prospective non-randomized clinical trial that will test the effectiveness of SCION-HSCT program against care as usual on perceived HRQoL of the patient and the adherence to care program.

Oncology patients with HSCT will be recruited by the nurses of the participating wards under the guidance of a research nurse. They will be included in the trial if they will meet the inclusion criteria and signed informed consent (the full inclusion criteria see below).

Groups will be treated consecutively. The first group will receive care as usual (Control). After finishing the control period, i.e. after 42 Patients will have completed the trial. The the newly assigned patients will be treated according to SCION-HSCT program a multi-modular somatic-psycho-social care intervention (Intervention).

The intervention will be conducted by specially trained ward nurses in cooperation with the research nurse. It includes components of knowledge, skills training, and coaching to improve patients adherence to self management strategies for physical activity, prevention of oral mucositis and mal nutrition prevention. The HRQoL, adherence and symptom level of the patients will be observed up to 100 days post HSCT. Both quantitative and qualitative analyses will be conducted to evaluate patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Hematologic Patients (> 14 years of age)
* Hematological stem cell transplantation (HSCT) allogenic or autologous
* Informed consent

Exclusion Criteria:

* Unable to read, write, and understand German

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2007-12; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Health Related Quality of Life (HRQoL) | day before discharge from hospital

SECONDARY OUTCOMES:
Physical Fitness (Step-Test) | day before discharge from hospital
Fatigue (Fatigue Symptom Inventory - D (German)) | day before discharge from hospital
Physical Resources (German Conservation of Resources Evaluation (GCOR)) | day before discharge from hospital
Symptom experience (Common Terminology Criteria for adverse events - CTCAE v. 3.0) | day before discharge from hospital

CONTACTS AND LOCATIONS:
Locations (1):
- Martin-Luther-University Halle-Wittenberg, Medical Faculty, Department for Health and Nursing Science, Halle, Saxony-Anhalt, Germany

REFERENCES:
- See also: Presentation (12.2007) for work group in psycho oncological cancer care — http://www.pso-ag.de/Beitraege07/Landenberger%20KMT-Projekt.pdf